CLINICAL TRIAL: NCT01150110
Title: Evaluation of Resilient Occlusal Splints in the Control of Patients With Temporomandibular Disorder (TMD)
Brief Title: Resilient Occlusal and Patients With Temporomandibular Disorder (TMD)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Purpose: Treatment
Other Study IDs: 432
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2007-05

CONDITIONS: Temporomandibular Disorders
Keywords: Temporomandibular disorders; occlusal splints; electromyography; TMD (muscle and joint dysfunction); masseteres e anterior temporalis muscles.
MeSH Terms: conditions — Temporomandibular Joint Disorders; Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: resilient occlusal splints — A resilient occlusal splints (silicone 2mm) was fabricated on the maxillary arch, using a vacuum pressing machine. The occlusal splints were adjusted to eliminate the gross interferences and to obtain occlusal stability with maximum posterior bilateral contacts.
  Patients were instructed to use the occlusal splints for 24 hours during 30 days. The use was interrupted only during meals.

SUMMARY:
The purpose of this study was to compare the effectiveness of soft occlusal splint therapy on the electromyographic activity of masticatory muscles (ateriors temporalis and masseter) before and after the application of a muscle relaxation splint. Electromyography recordings from the masseter and anterior temporalis muscles were analyzed quantitatively during maximal clench, rest and mastication usual, before and after the treatment without a splint. Ten patients whose chief complaint was Temporomandibular Disorders (TMD) were selected for the study. After the initial evaluations soft occlusal splints (muscle relaxation splints) were applied, and the patients were instructed to use the splints for four weeks. Surface electromyographic recordings were taken from each patient, as clinical evaluations of TMD (Index of Helkimo), both evaluations before the beginning of clinical therapy and after four weeks of wearing splints. The data obtained were analyzed by Wilcoxon´s and Friedman´s tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and/or diagnosis of TMD
* With complaints of muscle disorders and / or joint pain, pain symptoms
* Presence of occlusal interferences
* Minimum of 20 functional teeth in the oral cavity with subsequent bilateral occlusion

Exclusion Criteria:

* Individuals with extensive dental flaws
* Orthodontic treatment in progress
* History of systemic diseases as advanced arthritis, diabetes and conservative and reversible treatments such as occlusal splints are recommended

Ages: 19 Years to 50 Years | Sex: All
Age Groups: Adult
Dates: Start 2007-07; Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Germana Camargos, academic, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Germana De Villa camargos, Uberlândia, Minas Gerais, Brazil